CLINICAL TRIAL: NCT03697876
Title: Phase I Clinical Study, to Evaluate the Safety and Tolerability of the Ophthalmic Gel PRO-165 Versus Artelac® Nightime Gel, on the Ocular Surface of Ophthalmological and Clinically Healthy Subjects
Brief Title: Safety and Tolerability of the Ophthalmic Gel PRO-165 Versus Artelac® Nightime Gel
Acronym: PRO-165
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH165-0217/I
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Syndromes
Keywords: PRO-165; sodium hyaluronate; Chondroitin sulfate 0.18%
MeSH Terms: conditions — Dry Eye Syndromes | interventions — chondroitin sulfate, sodium hyaluronate drug combination; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: controlled, of parallel groups, double blind, randomized, exploratory
Who Masked: Participant, Investigator
Masking Description: The blinding will correspond to the research subject and the principal investigator. In addition, the statistical analysis will be carried out in a blinded manner for the partial and final analysis.
  The masking will be done by means of identical labels. Which, in accordance with current and applicable regulations, must contain at least:
  * Name, address and telephone number of the sponsor
  * Pharmaceutical form and route of administration
  * Lot Number
  * Legend "Exclusively for clinical studies"
  * Date of Expiry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-165 (Experimental): Dose: one drop of gel, 4 times a day during the waking period, in the bottom of the right eye sac
  Interventions: Drug: PRO-165
- 1. Artelac® Nightime Gel (Active Comparator): Dose: one drop of gel, 4 times a day during the waking period, in the bottom of the right eye sac

INTERVENTIONS:
Drug: PRO-165 — PRO-165 Chondroitin sulfate 0.18% / sodium hyaluronate 0.2%, ophthalmic gel. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
  Other Names: sodium hyaluronate 0.2%; chondroitin sulfate + sodium hyaluronate; chondroitin sulfate 0.18%
  Arms: PRO-165
Drug: Artelac — Artelac® Nightime Gel. 0.2% Carbomer, ophthalmic gel. Made in Germany by: Dr. Gerhard Mann Chem Pharm. Imported and marketed by: Bausch & Lomb México, S.A. de C.V.
  Other Names: Carbomer 0.2%

SUMMARY:
Objective: To assess the safety and tolerability of the PRO-165 formulation on the ocular surface of ophthalmologically and clinically healthy subjects.

Hypothesis: Ophthalmic gel PRO-165 presents a safety and tolerability profile similar to Artelac® Nightime Gel in ophthalmological and clinically healthy subjects.

Phase I clinical study, controlled, of parallel groups, double blind, randomized, exploratory Therapeutic indication of PRO-165: Eye lubricant

DETAILED DESCRIPTION:
The study subjects will be recruited from various research centers in western and central Mexico.

Each research center has a monitoring plan specified according to the recruitment capabilities of the same, which must be at least once a month, where the queries of your data entered into the electronic case report report will be reported to the center. (e-CRF) for which it has as time limit the next monitoring visit to make the pertinent changes.

The report of adverse events will be made according to the standard operating procedure (PNO) where it specifies, according to Official Mexican Standard 220 (NOM 220), that the signs or symptoms of adverse events will be reported based on the Medical Dictionary. for Regulatory Activities, for which the sponsor has version 20.1 in Spanish. For serious adverse events (SAEs) will be reported in accordance with the standardized operation procedure of pharmacovigilance of the sponsor, which adheres to the guidelines of NOM 220 and international regulations, these will be reported in the regulatory framework to the regulatory entity within a period of time no more than 7 days.

The study is registered in the National Registry of Clinical Trials (RNEC), entity equivalent to Clinical Trials in Mexico.

The quality assurance plan is carried out by the sponsor through the Quality Assurance agent in Clinical Research, whose function is to conduct inspections and audits of the research sites to document and generate reports of deviations from the protocol. In addition to the visits of the monitoring plan, the reliability of the data is guaranteed.

To verify the integrity, veracity and reliability of the data entered into the e-CRF, the monitors of each center will check the information uploaded to the portal with that reported in the source document of the principal investigator (PI), such as clinical notes, clinical history and documents. and formats attached to the research protocol, physical case report format, as well as those provided by the sponsor to the PI (subject's diary and quality and satisfaction survey).

The e-CRF used for this clinical study is provided by an internationally certified provider with the highest quality standards, protection of information under current regulations and confidentiality guarantee. The information that the PIs enter into the e-CRF is collated and verified by the clinical monitors and by the service provider's personnel, later reviewed and approved by the medical ophthalmologist researcher and by the Clinical Security Pharmacologist, who authorize the monitored data of clinical information and safety of the study molecule, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Systemically and ophthalmologically healthy subjects evaluated during the clinical history.
* Age between 18 to 45 years.
* Both genders.
* Blood tests (complete blood count, three element blood chemistry and liver function tests within normal parameters specified by the reference laboratory with a lower and upper margin of 10%)
* Vital signs within normal parameters. (Vital signs at rest: blood pressure ≤ 139/89 mmHg, heart rate 60 -100 beats per minute and respiratory rate of 12-24 breaths per minute)
* Visual capacity 20/30 or better, in both eyes.
* Intraocular pressure ≥11 and ≤ 21 mmHg.

Exclusion Criteria:

* Subjects with a history of hypersensitivity to any of the components of the research products.
* Subject users of topical ophthalmic medications of any pharmacological group.
* Subject users of medication by any other route of administration.
* Women who are pregnant or lactating.
* Women without a history of bilateral tubal obstruction, oophorectomy or hysterectomy, who do not ensure a hormonal contraceptive method or intrauterine device during the study period.
* Subjects with participation in clinical research studies 90 days prior to inclusion in the present study.
* Known diagnosis of liver disease
* Inability to attend or answer the evaluations made in each of the visits.
* Positive tobacco use (specified as cigarette consumption regardless of quantity and frequency)
* Positive alcoholism (specified as the consumption of alcoholic beverages, regardless of quantity and frequency, during the study intervention period).
* Contact lens users.

Medical and therapeutic exclusion criteria.

* History of any chronic-degenerative disease.
* Inflammatory or infectious disease, active at the time of study entry.
* Injuries or traumatisms not resolved at the time of entry into the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Leslie victoria Aguilar Saldaña, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The principal investigator must request the authorization of the sponsor in writing to disseminate or communicate any type of information about the investigation.

RESULTS

PARTICIPANT FLOW:
Groups:
- 1. Artelac® Nightime Gel: Dose: one drop of gel, 4 times a day during the waking period, in the bottom of the right eye sac
  Artelac: Artelac® Nightime Gel. 0.2% Carbomer, ophthalmic gel. Made in Germany by: Dr. Gerhard Mann Chem Pharm. Imported and marketed by: Bausch & Lomb México, S.A. de C.V.
Period: Overall Study
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Started | 16 | 16
Visit 1 (The intention-to-treat (ITT) population is defined as any subject who has received at least one dose of the investigational product and concluded at least visit 1, regardless of their adherence to product or protocol. In this group, one subject did not undergo the final visit evaluations, but did participate in visit 1, so was considered for the safety variables as part of the ITT population) | 16 | 15
Completed (The analysis of the primary outcome variables of safety and tolerability was carried out in the per protocol (PP) population, defined as all subjects with the required adherence, and who concluded their participation without deviations from the study protocol. In this group one subject did not complete the study but was considered in the ITT population since the V1 did take place.) | 15 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Clincally healthy adult volunteers. There were 16 subjects included in each group initially (n=32), however, one subject from the control group was lost to follow-up and did not attend to any visits beyond scrutiny, impossible to confirm if any exposure to the product happened, and was not considered in any analyses.One patient in the PRO-165 group was lost during the course of the study, but did attend to Visit 1, so this subject was included in the ITT population (31) but not in the PP (30).
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.81 (4.7) | 28.87 (8.7) | 27.29 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 16 | 15 | 31
Height [Mean (Standard Deviation); unit: meters] | 1.67 (0.1) | 1.66 (0.1) | 1.66 (0.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 67.19 (9.0) | 69.53 (12.3) | 68.32 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The Principal Investigator will register the Events Adverse (EA) that the subjects of the study will present. The EAs will be expressed as absent or present and the number of cases will be counted by study group.
Time Frame: Throughout the 13 days of evaluation, including the safety call (day 13).
Population: One patient in the PRO-165 group was lost during the course of the study, but did attend to Visit 1, so this subject was included in the ITT population, and therefore considered for the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 16 | 15
Participants | 3 | 5

2. Primary Outcome: Ocular Comfort Index
Description: It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100). A higher score is a worse outcome.
  Similar to the index for ocular surface diseases, the ocular comfort index (ICO) evaluates symptoms. The ICO contains 6 items that focus on the discomfort associated with the ocular surface. Each of these questions has two parts, which inquire separately the frequency and severity of the symptoms.
  The evaluator will deliver the questionnaire to the subject and allow the subject to answer it calmly without any pressure and / or coercion, will only assist him if he has difficulty understanding any of the questions.
Time Frame: Baseline Visit (day 0) and Final Visit (day 11)
Population: The PP population was considered for this variable's data analysis. One patient in the PRO-165 group was lost during the course of the study, but did attend to Visit 1, so this subject was included in the ITT population (31) but not in the PP (30).
Measure: Mean (Standard Deviation); unit: Scores in a Scale
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 15 | 15
Scores in a Scale
  Baseline Visit (day 0) | 20.36 (13.3) | 15.37 (14.1)
  Final Visit (day 11) | 15.47 (11.9) | 10.99 (12.8)

3. Secondary Outcome: Visual Acuity (VA)
Description: Visual acuity (VA) is a test of visual function. It will be evaluated without refractive correction with the Snellen chart. The Snellen chart is the standard tool used to evaluate visual acuity. It was located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated. The contralateral eye to which it will be evaluated is covered, then the examiner detects until the line can clearly see the letters given he or she a score, the normal score for a VA is 20/20.This score can be expressed in both fraction (i.e. 20/20) or decimal (i.e. 0.5) formats. In this study, VA is expressed in fraction format.
Time Frame: Baseline Visit (day 0), Visit 1 (day 5), and Final Visit (day 11)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Decimal Score (Snellen Chart)
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 15 | 15
Decimal Score (Snellen Chart)
  Baseline Visit (day 0) | 19.33 (3.7) | 18.00 (2.5)
  Visit 1 (day 5) | 19.33 (3.7) | 19.33 (3.7)
  Final Visit (day 11) | 20.00 (4.6) | 18.67 (4.0)

4. Secondary Outcome: Intraocular Pressure (IOP)
Description: Tonometry is the objective measure of Intraocular pressure, based primarily on the force required to flatten the cornea, or the degree of corneal indentation produced by a fixed force. Goldman's tonometry is based on the Imbert-Fick principle. the result will be expressed in millimeters of mercury and the comparison between groups will be carried out.
Time Frame: Baseline Visit (day 0), Visit 1 (day 5), and Final Visit (day 11).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 15 | 15
mmHg
  Baseline Visit (day 0) | 14.13 (2.8) | 14.20 (3.6)
  Visit 1 (day 5) | 13.73 (2.5) | 13.53 (2.8)
  Final Visit (day 11) | 13.83 (2.5) | 14.00 (2.6)

5. Secondary Outcome: Number of Participants With Post-instillation Symptomatology
Description: The subject will be questioned if after applying the medication he felt burning, pruritus, a foreign body sensation and blurred vision.
  Presence or absence: it will be marked as present (1) or absent (0) for each of the symptoms questioned
Time Frame: Final Visit (day 11)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 15 | 15
Participants
  Burning sensation | 4 | 8
  Pruitus | 7 | 6
  Foreign Body Sensation | 9 | 8
  Blurry Vision | 15 | 15

6. Secondary Outcome: Tear Breakup Time (TBUT)
Description: Tear Breakup Time (TBUT) is a continuous variable that will be measured in seconds, evaluating the time it takes to break it, is done by direct counting and the normality range and mayor to 10 seconds.
Time Frame: Baseline Visit (day 0), Visit 1 (day 5), and Final Visit (day 11).
Population: One patient in the PRO-165 group was lost during the course of the study, but did attend to Visit 1, so this subject was included in the ITT population (31) but not in the PP (30). The PP population was considered for this variable's data analysis.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 15 | 15
Seconds
  Baseline Visit (day 0) | 12.67 (2.9) | 12.80 (3.0)
  Visit 1 (day 5) | 13.53 (3.4) | 13.47 (3.1)
  Final Visit (day 11) | 13.47 (3.9) | 13.40 (2.8)

7. Secondary Outcome: Number of Participants With Epithelial Defects (ED; Graded According to Oxford Scale)
Description: The epithelial defects will be evaluated by means of two stains, lysamine green and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the Oxford Scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects. The outcome describes the number of pariticipants who presented which grade according to the Oxford Scale.
Time Frame: Baseline Visit (day 0), Visit 1 (day 5), and Final Visit (day 11).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
Number analyzed (Participants) | 15 | 15
Participants
  Lysamine Green Day 0 (Basal Visit): Grade 0 | 15 | 15
  Lysamine Green Day 0 (Basal Visit): Grade 1 | 0 | 0
  Lysamine Green; Visit 1 (day 5): Grade 0 | 15 | 15
  Lysamine Green; Visit 1 (day 5): Grade 1 | 0 | 0
  Lysamine Green; Final Visit (day 11): Grade 0 | 15 | 15
  Lysamine Green; Final Visit (day 11): Grade 1 | 0 | 0
  Fluorescein; Baseline Visit (day 0): Grade 0 | 15 | 14
  Fluorescein; Baseline Visit (day 0): Grade 1 | 0 | 1
  Fluorescein; Visit 1 (day 5): Grade 0 | 15 | 15
  Fluorescein; Visit 1 (day 5): Grade 1 | 0 | 0
  Fluorescein; Final Visit (day 11): Grade 0 | 15 | 14
  Fluorescein; Final Visit (day 11): Grade 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected until day 13±1 of the study
Description: The Adverse Event Report considered the Intention-To-Treat (ITT) population, (16 for PRO-165 and 15 for Artelac® Nightime Gel; 31 total) all participants who were randomized and exposed to treatment (even one dose). There was one subject from the Artelac® Nightime Gel group who was lost to follow-up and did not attend to any visits beyond scrutiny, so it was impossible to confirm if any exposure to the product had taken place, and therefore not considered in the report.
Arm/Group | PRO-165 | 1. Artelac® Nightime Gel
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 3/16 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-165 (N=16) | 1. Artelac® Nightime Gel (N=15)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Iriitation in instillation site (Eye disorders) | 0 (0) | 5 (5)
Instillation site lacrimtion (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Admisnistration site pruritus (Eye disorders) | 0 (0) | 2 (2)
Eosinophil count Abnormal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Instillation site foreign body sensation (Eye disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT03697876/Prot_001.pdf
  • Statistical Analysis Plan (2017-07-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT03697876/SAP_002.pdf